CLINICAL TRIAL: NCT03224689
Title: A Multi-Centre Clinical Investigation To Evaluate The Safety And Performance Of The Freedom Total Knee® System With The PEEK-OPTIMA Femoral Component
Brief Title: Evaluation of The Safety And Performance of The Freedom Total Knee® System With The PEEK-OPTIMA Femoral Component
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maxx Orthopedics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MI-001
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Osteoarthritis, Knee; Rheumatoid Arthritis of Knee; Traumatic Arthritis of Knee (Diagnosis); Polyarthritis; Fractures, Bone
MeSH Terms: conditions — Osteoarthritis, Knee; Disease; Arthritis; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEEK Femoral (Experimental): Subjects with a primary diagnosis of end-stage symptomatic primary knee osteoarthritis who require a uni-lateral knee prosthesis and have been evaluated as appropriate candidates for a total knee arthroplasty by the Investigator will be invited to take part in this clinical investigation.
  Interventions: Device: PEEK-Optima Femoral Component

INTERVENTIONS:
Device: PEEK-Optima Femoral Component — TKA Surgery

SUMMARY:
Prospective, multi-centre, non-comparative, post-market surveillance clinical study

DETAILED DESCRIPTION:
PRIMARY ENDPOINT:

* The primary endpoint is to evaluate the procedural success ie successful implantation of the device in the opinion of the surgeon

SECONDARY ENDPOINTS:

The secondary endpoints are to evaluate:

* KSS Knee scores and KSS Function scores at 6 weeks, 6, 12 and 24 months post-treatment compared to pre-treatment
* Subject reported outcomes (SF-36, Oxford Knee Score and WOMAC) at 6 weeks, 6, 12 and 24 months post-treatment compared to pre-treatment
* Stability of the device through radiographic analysis to assess alignment and component position at immediate post-treatment, 6 weeks, 6, 12 and 24 months post-treatment
* Safety in terms of adverse events and device deficiencies throughout the clinical investigation including any additional knee treatments and/or surgery
* Survivorship analysis of the device at 12 and 24 months and annually thereafter

ELIGIBILITY:
INCLUSION CRITERIA:

* Male and female subjects aged 50 years of age or older and less than 75 years of age (>50 and <75 years).
* Subjects who require a uni-lateral knee prosthesis and have been evaluated as appropriate candidates for a total knee arthroplasty by the Investigator.
* Subjects with a primary diagnosis of end-stage symptomatic primary knee osteoarthritis
* Subjects who, in the opinion of the Investigator, are able to understand this clinical investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.
* Subjects who are able to give voluntary, written informed consent to participate in this clinical investigation and from whom consent has been obtained.

EXCLUSION CRITERIA:

* Subjects who, in the opinion of the Investigator, have an existing condition that would compromise their participation and follow-up in this clinical investigation.
* Subjects who are known drug or alcohol abusers or with psychological disorders that could affect follow-up care or treatment outcomes.
* Subjects who have participated in a clinical study with an investigational product in the last 6 months.
* Subjects with other significant disabling problems from the muscular-skeletal system other than in the knees (i.e muscular dystrophy, polio, neuropathic joints).
* Subjects with a BMI of 32 or above.
* Subjects with a current or active history of malignancy, active or suspected infection, Paget's disease, renal osteodystrophy, immunologically suppressed, rheumatoid arthritis, sickle cell anemia, and systemic lupus erythematosus.
* Subjects with a primary or secondary diagnosis of inflammatory or traumatic arthritis.
* Subjects defined by the Investigator as ASA Grade III or IV.
* Subjects who have a neuromuscular or neurosensory deficit.
* Female subjects who are pregnant or lactating.
* Subjects with an anatomical limb alignment of above 20 degrees varus or valgus.
* Subjects with a fixed flexion deformity of over 20 degrees.
* Subjects with recurvatum (definition: hyperextension ≥ 5 degrees).
* Subjects who have previously undergone total or unicondylar knee arthroplasty, high tibial osteotomy, ligament reconstruction, ORIF or with previous fracture in the ipsilateral knee joint.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Knee Society Score (KSS) | Change from Pre-op versus 6 weeks, 3 months, 6 months,12 months and 24 months
  Pre-and post-operative function and patient and mechanical assessment. The KSS contains questions in 2 sections: knee joint (pain, range of motion, stability) and function (walking distance, ability to climb stairs). The greater score correlates to better outcome.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | Change from Pre-op versus 6 weeks, 3 months, 6 months,12 months and 24 months
  Patient self administered overall satisfaction (scale from 1 worse -10 best)
SF-36 | Change from Pre-op versus 6 weeks, 3 months, 6 months,12 months and 24 months
  Assessment domains to explain variations in patient outcomes. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | Change from Pre-op versus 6 weeks, 3 months, 6 months,12 months and 24 months
  Assessment of OA of the knee or hip. Possible score range of 0- 20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function
Radiographic assessment | Change from Pre-op versus 6 weeks, 3 months, 6 months,12 months and 24 months
  Subjective review and assessment of serial radiographs. Items include presence or absence of radiographic evidence of component loosening, malposition, migration and periprosthetic osteolysis, bone loss or interface composite (bone-cement-component) breakdown.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Verdonk, MD, PhD, Principal Investigator — More Institute, Antwerp, Belgium
Locations (1):
- More Institue, Department of Orthopedic Surgery, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No